CLINICAL TRIAL: NCT00471575
Title: Prospective Observational Study
Brief Title: Fatty Liver in Pregnancy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Other Study IDs: 38/07
Record Dates: First submitted 2007-05-09; First posted 2007-05-10 (Estimated); Last update posted 2007-05-15 (Estimated); Status verified 2007-04

CONDITIONS: Fatty Liver
Keywords: fatty liver; pregnancy; ultra sound; Pregnant women at the end of pregnancy or immediately after birth.; controls-women with normal liver; correlation between ultrasonography and nutritional, obsthetric and laboratory data.
MeSH Terms: conditions — Fatty Liver

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: ultra sound examination

SUMMARY:
Non alcoholic fatty liver disease (NAFLD) is one of the main causes of development of chronic liver disease and cirrhosis. There are no published studies which have investigated the incidence of NAFLD in pregnant women or the correlation between the metabolic changes in pregnancy and this phenomenon.

We aimed in our study to explore the incidence of NAFLD in pregnancy by ultrasonography (US) during the end of the pregnancy or immediately after birth (after 36 weeks) and to look for a correlation between fatty liver and demographic, clinical, nutritional and laboratory data during pregnancy.

DETAILED DESCRIPTION:
Fatty liver in pregnancy-protocol:

Non alcoholic fatty liver disease (NAFLD) is one of the main causes of development of chronic liver disease and cirrhosis. The incidence of NAFLD among the general population is about 17-30%. There are no published studies which have investigated the incidence of NAFLD in pregnant women or the correlation between the metabolic changes in pregnancy and this phenomenon.

We aimed in our study to explore the incidence of NAFLD in pregnancy by ultrasonography (US) during the end of the pregnancy or immediately after birth (after 36 weeks) and to look for a correlation between fatty liver and demographic, clinical, nutritional and laboratory data during pregnancy.

Methods: US examination will be performed by an experienced technician. The liver will be scanned by B mode US using a 2-5 MHZ transducer. In those with fatty liver as seen by US, a repeat examination will be performed after 6 weeks and 24 weeks. For women with the diagnosis of fatty liver, serum lipid profile, glucose, liver function tests and insulin will be done. Homa score as well as BMI will be calculated for each woman with fatty liver. All participants will sign an informed consent which has been approved by the hospital ethical committee.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women during the end of the pregnancy or immediately after birth (after 36 weeks)

Exclusion Criteria:

* Pregnant women before 36 weeks of pregnancy.
* Known diabetes or treatment by drugs known to cause fatty liver.

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Dates: Start 2007-06; Study Completion 2007-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: efrat Broide, MD, Principal Investigator — Ethic committee of Assaf Harofeh Medical Center
Locations (1):
- Assaf Harofeh Medical Center, Ẕerifin, Israel